CLINICAL TRIAL: NCT01037205
Title: Randomized, Double-blind, Placebo Controlled Phase II Study to Examine the Effects of DAS181 in Healthy Adult Subjects With Laboratory Confirmed Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ansun Biopharma, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAS181 - 2 - 03 (DMID 09-0090); HHSN266200600015C (Other Grant/Funding Number: DMID)
Record Dates: First submitted 2009-12-18; First posted 2009-12-22 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2013-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DAS181 High Dose (Active Comparator): DAS181 Dry Powder 10 mg qd x 3 days
  Interventions: Drug: DAS181 dry powder, formulation F02
- DAS181 Low Dose (Active Comparator): DAS181 Dry Powder 10 mg Day 1 Lactose Placebo Day 2 and Day 3
  Interventions: Drug: DAS181 dry powder, formulation F02
- Lactose Placebo (Placebo Comparator): Lactose (Respitose ML006 (DMV-Fonterra)) 1 capsule qd x 3 days
  Interventions: Drug: Respitose ML006 (DMV-Fonterra)

INTERVENTIONS:
Drug: DAS181 dry powder, formulation F02 — 10 mg delivered dose DAS181 in clear HPMC #3 Capsules
  Arms: DAS181 High Dose; DAS181 Low Dose
Drug: Respitose ML006 (DMV-Fonterra) — Lactose monohydrate
  Arms: Lactose Placebo

SUMMARY:
This protocol will seek to enroll adult otherwise healthy subjects presenting with influenza-like illness (ILI). Subjects will enter the study based on listed inclusion/exclusion criteria, including a positive diagnostic test for influenza virus (IFV).

DETAILED DESCRIPTION:
This protocol will seek to enroll adult otherwise healthy subjects presenting with influenza-like illness (ILI). Subjects will enter the study based on listed inclusion/exclusion criteria, including a positive diagnostic test for influenza virus (IFV).

Based upon a Rapid Diagnostic Test of IFV, subjects will be randomized into one of three groups: a single dose DAS181 10 mg group, a multiple dose DAS181 10 mg, 10 mg, 10 mg dose group or a placebo group.

The full analysis set will include subjects with confirmed influenza as documented with Rapid Diagnostic Testing. The set will be used for activity analysis and will include all randomized subjects with baseline and treatment data. Study staff may visit subjects outside the clinic. Per protocol, the safety analysis sets are described below in Statistical Methods.

Peripheral venous blood samples for pharmacokinetic (PK) and immunogenic analysis of DAS181 will be obtained on 10 subjects enrolled in each study arm.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects in generally good health in the opinion of the investigator as determined by vital signs, medical history, and a targeted physical exam based on medical history.
2. Subjects must be able to verbalize understanding of the consent form, provide written informed consent and verbalize willingness to complete study procedures.
3. Be 18 to 70 years of age (inclusive).
4. Subjects must weigh at least 55 kg and must have a Body Mass Index (BMI) of no greater than 35.99
5. Febrile, oral temperature >100°F (37.8°C) and one or more of the following:

   * Respiratory symptom (cough, sore throat, nasal symptoms)
   * Constitutional symptom (headache, myalgia, sweat/chills, prostration)
6. Positive rapid antigen test (RAT) for influenza performed using FDA-Cleared and CLIA-Waived commercially available rapid antigen test. A subject may be enrolled following a positive RAT of any manufacturer. Test may be conducted by a primary care physician prior to study enrollment if documentation of a positive RAT can be provided (documentation may consist of subjects medical records and must be included in subject documentation). A subject with a negative RAT result may still enroll if the sponsor and investigator agree that there is a known influenza outbreak circulating in the community. Blood pressure within normal limits (systolic 90-150 mmHg; diastolic 50-95 mmHg) and heart rate between 45 and 140 beats per minute.
7. Blood pressure within normal limits (systolic 90-150 mmHg; diastolic 50-95 mmHg) and heart rate between 45 and 140 beats per minute.
8. Onset of illness no more than 48 hours prior to diagnosis. Note: Time of onset of illness is defined as either (1) the time when the temperature was first measured as elevated (at least one degree (°C) of elevation temperature), OR (2) the time when the subject experienced the presence of at least one respiratory symptom or the presence of at least one constitutional symptom.
9. Female subjects must be post-menopausal (one year or greater without menses), surgically incapable of childbearing, practicing abstinence or practicing two effective methods of birth control. Acceptable methods may include intrauterine device, spermicide, barrier and hormonal contraception. A female subject must agree to practice an acceptable method of birth control during study period and for 12 weeks after study terminates. All female subjects regardless of menopausal status or surgical history must have had a negative urine pregnancy test (urine betahuman chorionic gonadotropin [hCG]) during the screening visit. The urine pregnancy test must be sensitive to at least 50 mU/mL of beta-hCG.
10. Male subjects must agree to use a medically accepted form of contraception from time of enrollment to 12 weeks after study termination.

Exclusion:

1. Have received any investigational drug or vaccine within 8 weeks prior to study drug dosing.
2. Have had a serious adverse reaction or hypersensitivity to any drug.
3. Have received blood products within 6 months of study enrollment.
4. Have concurrent cystic fibrosis, emphysema or previous episodes of anaphylaxis.
5. Have sickle-cell disease.
6. Allergy or history of allergy to milk or lactose.
7. Any history of congenital or acquired bleeding abnormalities.
8. Existence of any surgical, medical, or laboratory condition that, in the judgment of the clinical investigator, might interfere with the safety, distribution, metabolism or excretion of the drug.
9. Use of antiviral influenza medications within 10 days prior to screening (subjects will be prohibited from taking antiviral influenza medications during the course of the trial).
10. Current clinical evidence of a recognized or suspected uncontrolled non-influenza infectious illness with onset prior to screening.
11. Known hypersensitivity to DAS181.
12. Women who are pregnant (urine pregnancy test), who are attempting to become pregnant, or who are breast-feeding.
13. Uncontrolled seizure disorder or history of seizure activity within 12 months prior to study participation.
14. Any significant findings in the subject's medical history or physical examination that, in the opinion of the investigator, would affect subject safety or compliance with the dosing schedule.
15. Documented infection other than IFV in past 2 weeks.
16. Subjects with previous or current history of asthma or COPD requiring acute or chronic medication.
17. Subjects with acute diagnosis of a chronic medical condition within the last 3 months.
18. Subjects with a chronic medical condition that have initiated or changed dosing or regimen of prescription medications for their chronic medical condition within the last 3 months (any changes in chronic medications during the 28 day enrollment period will be captured in the source documentation under concomitant medications).
19. Subjects with previous or current history of the following systemic disorders: immunological disorders, HBV, HCV or cirrhosis, transplant recipients, HIV infection, or other immunosuppressive illness.
20. Subjects with cancer or history of hematologic malignancy. Cancer is defined as any active neoplastic diseases excluding noninvasive basal cell carcinoma.
21. Subjects who have had or are scheduled to have surgery within 30 days of initiation of the study.
22. Subjects who have donated or lost more than 500 mL of blood in the two months prior to screening.
23. Psychiatric or cognitive illness or recreational drug/alcohol use that, in the opinion of the principal investigator, would affect subject safety and/or compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Level of influenza viral load as Area Under the Curve at Day 5 (AUC0 d5) as measured by a) quantitative polymerase chain reaction (quantitative PCR) and b) 50% tissue culture infectious dose (TCID50) in cell culture | 28 days
Safety and toxicity profile: Unacceptable Serious Adverse Events | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Moss, MD, Study Director — Ansun Biopharma, Inc.
Locations (42):
- United States (42):
  - Carmichael, California
  - Chula Vista, California
  - La Mesa, California
  - Lincoln, California
  - Los Angeles, California
  - Orange, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Hialeah, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Covington, Louisiana
  - Silver Spring, Maryland
  - North Dartmouth, Massachusetts
  - Bellevue, Nebraska
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Stony Brook, New York
  - Canton, Ohio
  - Dayton, Ohio
  - Franklin, Ohio
  - Groveport, Ohio
  - Miamisburg, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Ashland, Oregon
  - Lansdale, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Myrtle Beach, South Carolina
  - Simpsonville, South Carolina
  - Rapid City, South Dakota
  - Johnson City, Tennessee
  - Austin, Texas
  - Georgetown, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - West Point, Utah
  - West Valley City, Utah
  - Richmond, Virginia

REFERENCES:
- [Derived] Moss RB, Hansen C, Sanders RL, Hawley S, Li T, Steigbigel RT. A phase II study of DAS181, a novel host directed antiviral for the treatment of influenza infection. J Infect Dis. 2012 Dec 15;206(12):1844-51. doi: 10.1093/infdis/jis622. Epub 2012 Oct 8. PMID 23045618